CLINICAL TRIAL: NCT00889395
Title: Cognitive and Psychosocial Benefits of Caregiver Training for Ugandan HIV Children
Brief Title: Cognitive and Psychosocial Benefits of MISC Training for Ugandan Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Robert Opika Opoka, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R34MH082663-02 (NIH); 5R34MH082663-02 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-04

CONDITIONS: HIV; HIV Infections
Keywords: MISC; caregivers; children; psychosocial gains; cognitive benefits
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home visit (No Intervention): Patients will have monthly home visits during which health educational talks will be given
  Interventions: Behavioral: MISC training for primary caregivers

INTERVENTIONS:
Behavioral: MISC training for primary caregivers — Caregivers of children in the intervention arm will undergo a year long training in MISC
  Other Names: MISC group

SUMMARY:
The Mediational Interventions for Sensitizing Caregivers (MISC) model developed by Professor Pnina Klein is to enhance the cognitive and social development of children throughout the developing world . Although MISC has proven effective in a longitudinal study in two poorer communities of Addis Ababa, Ethiopia , it has not been used with HIV households or in the Ugandan context where there is desperate need for enhanced caregiving in HIV-affected families. We propose to work with community leaders, healthcare workers, and parents/caregivers in adapting MISC to the Ugandan cultural and social context in Kayunga. For intervention families, MISC training will be added to an ongoing home health care visit (HHCV) program already in place for HIV children in Kayunga district. We will then evaluate whether MISC parent/caregiver training improves cognitive and psychosocial development in their children, and whether clinical stability of the HIV child is an important modifier for MISC training benefit.

DETAILED DESCRIPTION:
In Uganda, about 110,000 children 0 to 14 years are living with AIDS however enhanced access to ARV medications has changed the prognosis for infected children from a uniformly deadly disease early in childhood to one in which survival well into adolescence is not uncommon. However, these prognostic changes have made psychosocial, educational, and quality-of-life considerations for the HIV child all the more critical. Studies on Ugandan HIV infected children show that they have cognitive, motor and emotional problems. These findings support the need for caregiving interventions with HIV children that extend beyond provision for basic medical and nutritional care only. These findings support the urgent need for programs that minister to the emotional and psychosocial needs of HIV-affected children.

The MISC is one such intervention that has proven effective in improving the cognitive, psychosocial and emotional needs of disadvantaged children. The MISC intervention is based on the use of naturally occurring situations and objects in the home environment. The process of training the caregivers in MISC theory and strategies is structured, whereas the process of implementing MISC with the children in the household is individualized and unstructured. The training of the caregiver is focused on the acquisition of knowledge and skills necessary for effective intervention to enrich the child's home-based learning environment.

Specific Objectives.

1. To establish the feasibility of MISC for caregivers of HIV infected children in Kayunga.
2. To investigate whether cognition and psychosocial functioning of HIV infected children are improved by MISC.
3. To determine whether cognitive and psychosocial gains for children of MISC-trained caregivers is moderated by disease severity of the child.

3. METHODS Phase 1: Adaptation of the MISC Study design. Adaptation of the MISC will be done using a cross sectional descriptive study. Prior to recruitment of participants, Prof. Klein will hold a series of focus group discussions (FDGs) in Kayunga to critique the MISC intervention.

Study population. Community leaders, health workers and parents/caregivers in Kayunga district, three FGDs will be held for each of these groups. They will partner with Dr. Klein in revising and adapting the MISC curriculum for training the local MISC staff who will accompany the CAI teams as they visit the HIV children and caregivers for the home health care visitation (HHCV). These CAI nursing staff will then train the caregivers each month as part of these HHCV visits.

Phase 2: MISC intervention Study design. This will be a randomized control study where HIV infected children younger than 6 yrs of age will be recruited and randomly assigned to either MISC intervention or non- intervention. All children will be recruited from the Child Health Advocacy International (CAI) project in Kayunga district during their routine home visits. Consecutive sampling will be used till the sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV positive children (ELISA and Western blot), less than six years of age.

Principal caregiver(s) of the eligible study child is able and willing to attend an initial daylong training session at a central location in Kayunga, followed by home-based monthly HHCV/MISC or HHCV support/training sessions for a one-year period and accompanying caregiving, as well as clinical/medical, cognitive, and psychosocial assessments for the child.

Exclusion Criteria:

* Medical history of serious birth complications or other known brain injury or disorder requiring hospitalization or continued evidence of seizure or other neurological disability.

Six years of age or older at start of study enrolled or planning to enroll in P1 (1st grade) level of school during the first 8 months of the year long intervention period.

Ages: 16 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes are children's cognitive and psychosocial assessment gains after year-long MISC training for their primary caregivers. | one year after commencement of MISC training

SECONDARY OUTCOMES:
Secondary outcomes are improved caregiving as a result of year long MISC training of caregivers. | one year after commencement of MISC training

CONTACTS AND LOCATIONS:
Overall Officials: Noeline Nakasujja, MD, Principal Investigator — Makerere University; Michael Boivin, PhD, Study Director — Michigan State University
Locations (1):
- Makerere University School of Health Sciences, Kampala, Uganda

REFERENCES:
- [Derived] Ikekwere J, Ucheagwu V, Familiar-Lopez I, Sikorskii A, Awadu J, Ojuka JC, Givon D, Shohet C, Giordani B, Boivin MJ. Attention Test Improvements from a Cluster Randomized Controlled Trial of Caregiver Training for HIV-Exposed/Uninfected Ugandan Preschool Children. J Pediatr. 2021 Aug;235:226-232. doi: 10.1016/j.jpeds.2021.03.064. Epub 2021 Apr 2. PMID 33819464
- [Derived] Ruisenor-Escudero H, Familiar-Lopez I, Sikorskii A, Jambulingam N, Nakasujja N, Opoka R, Bass J, Boivin M. Nutritional and Immunological Correlates of Memory and Neurocognitive Development Among HIV-Infected Children Living in Kayunga, Uganda. J Acquir Immune Defic Syndr. 2016 Apr 15;71(5):522-9. doi: 10.1097/QAI.0000000000000905. PMID 26605506
- [Derived] Boivin MJ, Bangirana P, Nakasujja N, Page CF, Shohet C, Givon D, Bass JK, Opoka RO, Klein PS. A year-long caregiver training program improves cognition in preschool Ugandan children with human immunodeficiency virus. J Pediatr. 2013 Nov;163(5):1409-16.e1-5. doi: 10.1016/j.jpeds.2013.06.055. Epub 2013 Aug 16. PMID 23958115